CLINICAL TRIAL: NCT04974762
Title: Comparing Truncal Blocks Versus Wound Infiltration for Subcutaneous Implantable Cardioverter Defibrillator Implantation
Brief Title: Truncal Blocks Versus Wound Infiltration for SICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ali Nima Shariat, Assistant Professor, Anesthesiology, Perioperative & Pain Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18-00379
Record Dates: First submitted 2021-07-08; First posted 2021-07-23 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Intraoperative Pain; Postoperative Pain
Keywords: Subcutaneous implantable cardioverter-defibrillators (S-ICD); Truncal blocks
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Masking Description: The researcher assessing the subjects postoperatively will be different from the anesthesiologist that performs the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound infiltration (Active Comparator): Standard intervention - surgical infiltration with local anesthetics
  Interventions: Procedure: Wound infiltration
- Truncal blocks (Experimental): Truncal block for anesthetics
  Interventions: Procedure: Truncal blocks

INTERVENTIONS:
Procedure: Wound infiltration — Surgical wound infiltration by proceduralist
  Arms: Wound infiltration
Procedure: Truncal blocks — Truncal blocks provided by anesthesiology team for device placement
  Arms: Truncal blocks

SUMMARY:
This is a single-center, randomized and prospective trial of all patients undergoing S-ICD implantation. Subjects will only be eligible for this study if they are ≥ 18 years of age and eligible to undergo S-ICD implant at Mount Sinai Morningside Hospital. They will be randomized to receive either surgical infiltration of local anesthetic or truncal blocks. Intraoperative and postoperative data will be collected including total opioid use, pain scores postprocedure, total postoperative narcotic need and length of stay.

DETAILED DESCRIPTION:
This is a single-center, randomized and prospective trial of all patients undergoing S-ICD implantation. Subjects will only be eligible for this study if they are ≥ 18 years of age and eligible to undergo S-ICD implant at Mount Sinai Morningside Hospital. They will be randomized to receive either surgical infiltration of local anesthetic or truncal blocks. Intraoperative and postoperative data will be collected including total opioid use, pain scores postprocedure, total postoperative narcotic need and length of stay. The procedures involved for the study are the placement of the described truncal blocks or wound infiltration. Data to be collected are patient demographics, history of present illness, past medical history, and pain management techniques required (i.e non-narcotics and narcotics use). In addition, age, race, gender and BMI will also be collected. Intraoperative analgesia requirements, postoperative analgesia requirements, duration of procedure and length of stay will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing S-ICD placement

Exclusion Criteria:

* Allergy to amide local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Intraoperative and postoperative opioid consumption | Up to Post-Op Day 10
  Total intraoperative and postoperative opioid consumption of subjects

SECONDARY OUTCOMES:
Non-opioid analgesic consumption | Up to Post-Op Day 10
  Total intraoperative and postoperative non-opioid analgesic consumption of subjects
Sedation (propofol) requirements intraoperatively | Day 1, Day of Surgery
  Total propofol required by subjects intraoperatively
Number of participants with ICU stay | Up to Post-Op Day 10
  Need of intensive care unit (ICU) stay
Duration of ICU stay | Up to Post-Op Day 10
  Duration of intensive care unit (ICU) stay
Visual Analog Pain score | Up to Post-Op Day 10
  Visual Analog Pain Score (VAS) - total scale from 0-10, with higher score indicating more pain
Total procedure time | Day 1 at Surgery
  Total duration of procedure time measured in minutes
Length of stay | Day 1 at Surgery
  Length of time in the postanesthesia care unit measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shariat, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Morningside Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).